CLINICAL TRIAL: NCT02781142
Title: The Effect of Telerehabilitation Based Motor Imagery Training on Gait and Balance Performance of the Persons With Multiple Sclerosis: A Randomized Controlled Trial
Brief Title: Motor Imagery Training in Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Turhan Kahraman, MSc, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2628-GOA
Record Dates: First submitted 2016-05-17; First posted 2016-05-24 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor imagery training (Experimental): Persons with multiple sclerosis
  Interventions: Other: Motor imagery training
- Control group (No Intervention): Persons with multiple sclerosis
- Healthy controls (No Intervention): Healthy participants

INTERVENTIONS:
Other: Motor imagery training — The motor imagery training will be designed for the individual basis with following standard protocols. It will be applied two times a week for 8 weeks. The first one and/or two sessions will be performed in the clinic, the other will be performed at the patients' home with a video-conference telerehabilitation technique.
  Arms: Motor imagery training

SUMMARY:
Motor imagery training facilitates the neural plasticity with increasing the neuronal cortical pathways in the brain. Motor imagery training is an effective way in stroke survivors. However, its effects in persons with multiple sclerosis (MS) are not known. Additionally, telerehabilitation based motor imagery training is very rare treatment way which requires more research. Therefore, this study aims to investigate the effect of telerehabilitation based motor imagery training on gait and balance performance of the persons with MS.

The participants will be allocated into three groups, including motor imagery training, wait-list control group, and healthy control group.

All the assessments will be performed before and after the training in the 8-week motor imagery training group. The participants in the control group will underwent the assessment with a 8-week interval. The healthy participants will be assessed only one.

The motor imagery training will be designed for the individual basis with following standard protocols. It will be applied two times a week for 8 weeks. The first one and/or two sessions will be performed in the clinic, the other will be performed at the patients' home with a video-conference telerehabilitation technique.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic, inflammatory, and demyelinating disease of the central nervous system. It is the most common neurological disease which causes progressive gait and balance disorders in young adults. The previous studies have indicated that home care and treatment services, which accelerates the healing process and makes the one feel better, are more preferred by the patients. Persons with MS are commonly not able to access the institutional rehabilitation services because of their disability and/or home location. It restricts the participation of the persons with MS and their treatment benefits. In recent years, the telerehabilitation programs are increasing to overcome this problem. Motor imagery training also stands as a good option in the rehabilitation programs. Motor imagery is a mental process by which an individual rehearses or simulates a given action. Motor imagery training facilitates the neural plasticity with increasing the neuronal cortical pathways in the brain. Motor imagery training is an effective way in stroke survivors. However, its effects in persons with MS are not known. Additionally, telerehabilitation based motor imagery training is very rare treatment way which requires more research.

The aim of this study is to investigate the effect of telerehabilitation based motor imagery training on gait and balance performance of the persons with MS.

The participants will be allocated into three groups, including motor imagery training group, control group, and healthy control group. The persons with MS will be recruited from the outpatient MS clinic of Dokuz Eylul University, and the healthy participants will be recruited from the stuff of Dokuz Eylul University.

The inclusion and exclusion criteria assessments and the neurological examination will be performed by a blinded neurologist specialized in MS. The cognition, fatigue, depression, and quality of life assessment will be performed by a blinded neuropsychologist. The remaining assessments, including walking, balance, and motor imagery abilities will be assessed by a blinded physiotherapist. All the assessments will be performed before and after the training in the 8-week motor imagery training group. The participants in the control group will underwent the assessment with a 8-week interval. The healthy participants will be assessed only one.

The motor imagery training will be designed for the individual basis with following standard protocols. It will be applied two times a week for 8 weeks. The first one and/or two sessions will be performed in the clinic, the other will be performed at the patients' home with a video-conference telerehabilitation technique.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis
* Having the Expanded Disability Status Scale 0 - 4.0
* Relapse-free period at the last 3 months
* Enough computer use ability
* Having computer and internet connection

Exclusion Criteria:

* Having severe musculoskeletal, cardiovascular, pulmonary, or metabolic disease
* Severe cognitive impairment
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Dynamic Gait Index | Change from Baseline at 8 weeks

SECONDARY OUTCOMES:
Expanded Disability Status Scale | At Baseline
Kinesthetic and Visual Imagery Questionnaire (KVIQ)-10 | Change from Baseline at 8 weeks
Movement Imagery Questionnaire-Revised Second Edition (MIQ-RS) | Change from Baseline at 8 weeks
Mental Chronometry for 2-Meter Walk Test | Change from Baseline at 8 weeks
Mental Chronometry for 5-Meter Walk Test | Change from Baseline at 8 weeks
Mental Chronometry for 10-Meter Walk Test | Change from Baseline at 8 weeks
Mental Chronometry for Timed 25-Foot Walk | Change from Baseline at 8 weeks
Mental Chronometry for Timed Up and Go Test | Change from Baseline at 8 weeks
Mental Chronometry for Five Times Sit to Stand Test | Change from Baseline at 8 weeks
2-Meter Walk Test | Change from Baseline at 8 weeks
5-Meter Walk Test | Change from Baseline at 8 weeks
10-Meter Walk Test | Change from Baseline at 8 weeks
Timed 25-Foot Walk | Change from Baseline at 8 weeks
2-Minute Walk Test | Change from Baseline at 8 weeks
Twelve Item MS Walking Scale | Change from Baseline at 8 weeks
Timed Up and Go Test | Change from Baseline at 8 weeks
Five Times Sit to Stand Test | Change from Baseline at 8 weeks
Curl-up Test | Change from Baseline at 8 weeks
Activities-specific Balance Confidence Scale | Change from Baseline at 8 weeks
Postural Stability Test by Balance System™ | Change from Baseline at 8 weeks
The Limits of Stability Test by Balance System™ | Change from Baseline at 8 weeks
Fall Risk Test by Balance System™ | Change from Baseline at 8 weeks
Modified Fatigue Impact Scale | Change from Baseline at 8 weeks
Hospital Anxiety and Depression Scale | Change from Baseline at 8 weeks
Multiple Sclerosis International Quality of Life Questionnaire | Change from Baseline at 8 weeks
Symbol Digit Modalities Test | Change from Baseline at 8 weeks
Selective Reminding Test | Change from Baseline at 8 weeks
10/36 Spatial Recall Test | Change from Baseline at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sema Savci, Prof, PhD, Study Director — Dokuz Eylul University; Turhan Kahraman, MSc, Principal Investigator — Dokuz Eylul University
Locations (2):
- Turkey (Türkiye) (2):
  - Dokuz Eylul University Hospital, MS Outpatient Clinic, Izmir
  - Dokuz Eylul University, School of Physical Therapy and Rehabilitation, Izmir

IPD SHARING:
Plan to Share IPD: Undecided